CLINICAL TRIAL: NCT02793440
Title: Clinical Results After Medical Therapy Alone or Medical Therapy Associated With Lumbar Traction in the Treatment of Nerve Root Pain of Lumbar Disc Herniation With Disco-radicular Conflict
Brief Title: Effectiveness of Lumbar Traction in Lumbar Disk Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO13106
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Lumbar Disk Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

ARMS (2):
- cortivazol (Active Comparator): anti-inflammatory therapy and epidural
  Interventions: Other: cortivazol treatment; Other: lumbar traction
- Traction arm (Experimental): Medical treatment associated with 5 lumbar traction sessions
  Interventions: Other: lumbar traction

INTERVENTIONS:
Other: cortivazol treatment
  Arms: cortivazol
Other: lumbar traction

SUMMARY:
The purpose of this study is to compare the clinical outcome of medical treatment associated with lumbar traction and medical treatment alone in the treatment of lumbar disk herniation.

DETAILED DESCRIPTION:
This is a prospective and randomized study. Medical treatment = anti-inflammatory therapy and epidural Medical treatment associated with lumbar traction medical treatment = + 5 lumbar traction sessions.

ELIGIBILITY:
Inclusion :

* patient with lumbar disc herniation with radiculopathy, over 18 years and consenting

Exclusion :

* sciatic complicated (motor deficit or cauda equina syndrome), against indication for medical treatment and / or lumbar traction
* previous lumbar surgery
* sciatica without disc herniation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2013-12-02 (Actual); Primary Completion 2022-07-02 (Estimated); Study Completion 2023-01-02 (Estimated)

PRIMARY OUTCOMES:
Decrease radicular pain (25%) | to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France